CLINICAL TRIAL: NCT04996485
Title: Scientific Substantiation and Assessment of the Effectiveness of Pathogenetic Methods of Therapy for Congenital Ichthyosis in Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Medical Research Center for Children's Health, Russian Federation (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12269723
Record Dates: First submitted 2021-07-21; First posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-07

CONDITIONS: Congenital Ichthyosis
Keywords: Congenital ichthyosis; Netherton syndrome; Autosomal recessive congenital ichthyosis; Biologic therapy
MeSH Terms: conditions — Ichthyosis Vulgaris; Netherton Syndrome | interventions — secukinumab; Ustekinumab; dupilumab

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Experimental group №1 (Secukinumab ) (Experimental): Secukinumab - subcutaneous injections into the shoulder according to the schedule of 0,1,2,3 weeks, then injections 1 time in 3 months up to 52 weeks of therapy.
  Interventions: Drug: Secukinumab Injection
- Experimental group №2 (Ustekinumab) (Experimental): Ustekinumab - subcutaneous injections in the shoulder on schedule 0; 1 month, then every 2 months up to 52 weeks of therapy.
  Interventions: Drug: Ustekinumab Injection
- Experimental group №3 (Dupilumab) (Experimental): Dupilumab - subcutaneous injections in the shoulder:
  for patients weighing from 15 to <30 kg: initial dose - 600 mg (2 injections of 300 mg), then 300 mg every 4 weeks; for patients weighing from 30 to <60 kg: initial dose - 400 mg (2 injections of 200 mg), then 200 mg every 2 weeks; for patients weighing 60 kg or more: the initial dose is 600 mg (2 injections of 300 mg), then 300 mg every 2 weeks.
  Interventions: Drug: Dupilumab Injection
- Control group (Symptomatic therapy) (Active Comparator): symptomatic therapy with emollients + systemic retinoids
  Interventions: Other: Symptomatic therapy

INTERVENTIONS:
Drug: Secukinumab Injection — Pathogenetic therapy with biologic drugs
  Arms: Experimental group №1 (Secukinumab )
Drug: Ustekinumab Injection — Pathogenetic therapy with biologic drugs
  Arms: Experimental group №2 (Ustekinumab)
Drug: Dupilumab Injection — Pathogenetic therapy with biologic drugs
  Arms: Experimental group №3 (Dupilumab)
Other: Symptomatic therapy — Active external agents, Emollients, systemic retinoids if needed
  Arms: Control group (Symptomatic therapy)

SUMMARY:
This is an experimental non-randomized clinical study aimed at expanding the indications for the use of biological drugs with the aim of using them for the pathogenetic therapy of children with congenital ichthyosis.

DETAILED DESCRIPTION:
This is an experimental non-randomized clinical study aimed at expanding the indications for the use of biological drugs with the aim of using them for the pathogenetic therapy of children with congenital ichthyosis.

The study will include 50 children aged 6 months to 18 years with a clinically and genetically confirmed diagnosis of congenital ichthyosis. Patients will be divided into 4 groups who will receive symptomatic therapy (using active external agents, emollients and / or systemic retinoids) or biologics targeting the cytokines IL-12 / IL-23, IL-4 / IL-13 and IL -17A. Immunophenotyping of all patients will be performed, the cytokine profile and spectrum of sensitization and the degree of NF-kB activation in lymphocytes will be determined. In experimental group №3, 10 patients with Netherton syndrome will receive dupilumab, in experimental group №2, 10 patients will receive ustekinumab, and in experimental group №1 10 patients will receive secukinumab. Efficiency will be assessed using the Ichthyosis Area Severity Index (IASI), determination of the level of TEWL, and the change in quality of life will also be assessed using the Children's Dermatological Life Quality Index (CDLQI) in comparison from baseline, than at 16 and 52 weeks. Throughout the study, the safety profile (registration of the development of infectious diseases) will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* The subject has signed an informed consent; parental or legal representative consent for patients under 18 years of age, as well as additional consent for patients aged ≥ 15 and <18.

  * At the time of participation in the study, the age of the subject is not less than 6 months and not more than 18 years.
  * At the time of participation in the study, a clinical diagnosis was established: Congenital ichthyosis with various clinical forms, with the exception of vulgar and X - linked congenital ichthyosis (genetic research is not a prerequisite for participation in the study).
* Subjects should have at least moderate IASI erythema associated with his / her ichthyosis, and a decrease in the quality of life according to CDLQI ≥ 10
* Absence of signs of severe infectious diseases (pneumonia, tuberculosis, etc.)
* No previous history of the use of the following genetically engineered biological drugs: ustekinumab, secukinumab, dupilumab

Exclusion Criteria:

* Subjects who have an allergic reaction to ustekinumab, secukinumab or other components of the drugs.
* Subjects who have bacterial and/or fungal diseases.
* Subjects who have problems in dynamic observation.
* Subjects who will have a worsening of clinical symptoms

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Ichthyosis Area Severity Index (IASI) | From Baseline up to 16 weeks
  Clinical measures included the Ichthyosis Area Severity Index (IASI), which integrates erythema (IASI-E) and scaling (IASI-S)
Change in Ichthyosis Area Severity Index (IASI) | 52 weeks
  Clinical measures included the Ichthyosis Area Severity Index (IASI), which integrates erythema (IASI-E) and scaling (IASI-S)

SECONDARY OUTCOMES:
Transepidermal water loss (TEWL) level change | From Baseline up to 16 weeks
  Change in transepidermal water loss (TEWL) while rebuilding the epidermal barrier of the skin (an indicator of the effectiveness of the therapy). Measured in g/hm2.
Transepidermal water loss (TEWL) level change | 52 weeks
  Change in transepidermal water loss (TEWL) while rebuilding the epidermal barrier of the skin (an indicator of the effectiveness of the therapy). Measured in g/hm2.
Change in the Children's Dermatology Life Quality Index (CDLQI) | From Baseline up to 16 weeks
  increasing The Children's Dermatology Life Quality Index, as an indicator of the effectiveness of therapy. The CDLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired. The CDLQI can also be expressed as a percentage of the maximum possible score of 30.
Change in the Children's Dermatology Life Quality Index (CDLQI) | 52 weeks
  Change in the Children's Dermatology Life Quality Index (CDLQI), as an indicator of the effectiveness of therapy. The CDLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired. The CDLQI can also be expressed as a percentage of the maximum possible score of 30.

CONTACTS AND LOCATIONS:
Locations (1):
- National Medical Research Center for Children's Health, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided